CLINICAL TRIAL: NCT03601312
Title: OC-Go: Facilitating Fidelity and Dissemination of Evidence Based Treatment for Childhood OCD Via an Interactive Crowd-sourced Patient-provider Tool
Brief Title: Randomized Controlled Trial of Standard ERP and OC-Go
Acronym: OC-GoPhaseII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Virtually Better, Inc. (Industry)
Responsible Party: Principal Investigator, John Piacentini, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R42MH111277-02 (NIH)
Record Dates: First submitted 2018-06-05; First posted 2018-07-26 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: All participants will receive 12 weeks of exposure/response/prevention (ERP). Sessions 1 (psychoeducation/hierarchy creation) and 12 (relapse prevention & generalization training) will be identical across both randomization groups.
  Treatment sequences for the randomization groups will be as follows:
  OC-GO-FIRST - Sessions 2-6: ERP+OC-Go, Sessions 7-11: Standard ERP
  STANDARD ERP-FIRST - Sessions 2-6: Standard ERP, Sessions 7-11: ERP+OC-Go
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not have information about the participant's treatment condition, so they will not know whether or not they are receiving treatment as usual (Standard ERP) or OC-Go augmented ERP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-As-Usual (Active Comparator): Individuals receiving treatment as usual will be receiving exposure and response prevention (ERP), the standard of care for pediatric OCD.
  Interventions: Behavioral: Exposure and Response Prevention
- OC-Go (Experimental): Individuals in the OC-Go group will be receiving exposure and response prevention (ERP) augmented by the OC-Go application.
  Interventions: Behavioral: OC-Go

INTERVENTIONS:
Behavioral: Exposure and Response Prevention — Exposure and response prevention is an evidence-based behavioral treatment that primarily focuses on exposures, in which the child faces OCD-related fears in a methodical manner and acquires more adaptive coping strategies.
  Arms: Treatment-As-Usual
Behavioral: OC-Go — OC-Go is a HIPAA-compliant web-based clinician portal and patient-side mobile application that allows clinicians to create and push tailored treatment assignments to patients on their mobile devices. Individuals receiving this intervention will receive exposure and response prevention with OC-Go.
  Arms: OC-Go

SUMMARY:
Phase II of this study will examine the efficacy of the OC-Go application via a randomized controlled trial comparing standard exposure and response prevention (ERP) treatment for pediatric obsessive compulsive disorder (OCD) to exposure/response prevention (ERP) augmented with OC-Go. A cross-over design will be implemented for these 12 sessions of treatment, in which participants that were randomized to standard ERP will receive OC-Go augmented ERP for the second half of treatment, and vice versa. Efficacy will be investigated in a sample of 32 children with OCD.

DETAILED DESCRIPTION:
This project seeks to refine and assess OC-Go, a HIPAA-compliant web-based clinician portal and patient-side mobile application designed to increase patient adherence to evidence-based treatment (EBT) for OCD, a common and impairing condition, and provider ability to effectively implement EBTs. OC-Go allows clinicians to create and push tailored assignments to patients on their mobile devices with an optimized user interface that includes patient accountability and support features. Accordingly, patients can be guided to do assignments by themselves between sessions with increased fidelity over the course of treatment. Once therapy assignments are created and shared to a crowd-sourced and curated public library, any clinician can assign any task to any patient for homework or in-session use with one touch. Use of OC-Go is expected to increase patient engagement, compliance, treatment efficiency, dissemination of EBTs, and therapist confidence and expertise.

ELIGIBILITY:
Inclusion Criteria:

* Ages 9-17 years old
* Primary diagnosis of OCD based on diagnostic interview (ADIS)
* CGI-Severity score > 3

Exclusion Criteria:

* Anti-OCD medication/unstable dose (with changes expected during the study)
* Significant and interfering comorbid psychiatric, psychosocial, neurological, or medical condition (e.g., acute suicidality, low IQ, etc.) precluding the child's ability to complete all study procedures

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Homework compliance | End of Week 14
  Homework Compliance (%; range 0-100) = (Total homework assignments completed treatment weeks 2-11/Total homework assignments assigned weeks 2-11) * 100

SECONDARY OUTCOMES:
Clinical Global Impression - Improvement Scale (acute) | End of Week 6
  The CGI-I is a single-item clinician-rated measure of global improvement. Scores range from 1 (very much improved) to 7 (very much worse), with scores of 1 or 2 (much improved) indicating positive treatment response.
Clinical Global Impression - Improvement Scale (crossover) | End of Week 14
  The CGI-I is a single-item clinician-rated measure of global improvement. Scores range from 1 (very much improved) to 7 (very much worse), with scores of 1 or 2 (much improved) indicating positive treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: John Piacentini, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Univ. of California / Los Angeles / Semel Inst., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No